CLINICAL TRIAL: NCT00687141
Title: A Phase I, Randomized, Double-blind (with-in Panel), Placebo-controlled, Parallel Group Study to Assess the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of AZD0328 in Healthy Elderly Volunteers After Oral Multiple Ascending Doses of AZD0328
Brief Title: Study to Assess the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of AZD0328 in Elderly Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Didier Meulien, M.D., Medical Science Director, Emerging Neuroscience, AstraZeneca Pharmaceuticals
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: D0190C00006; EudractCT 2007-004598-25
Record Dates: First submitted 2008-05-28; First posted 2008-05-30 (Estimated); Last update posted 2010-12-10 (Estimated); Status verified 2008-07

CONDITIONS: Alzheimer's Disease
Keywords: Safety; tolerability; AZD0328
MeSH Terms: conditions — Alzheimer Disease | interventions — spiro(1-azabicyclo(2.2.2)octane-3,2'(3H)-furo(2,3-b)pyridine)

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: AZD0328
- 2 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AZD0328 — Oral solution administered orally once per day on day 1, and then day 3 through to day 14. Specific dose depends on dose panel.
  Arms: 1
Drug: Placebo — Administered orally as a solution once per day on day 1, and then day 3 through to day 14.
  Arms: 2

SUMMARY:
The primary purpose of this study is to investigate the safety and tolerability of AZD0328 following once-daily dosing for 13 days in elderly healthy volunteers and to define maximum tolerated dose.

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed informed consent
* Clinically normal physical findings, laboratory values, vital signs and resting ECG as judged by the investigator

Exclusion Criteria:

* History of clinically significant cardio- or cerebrovascular, pulmonary, renal, hepatic, neurological, mental or gastrointestinal disorder or any other major disorder
* History of severe allergy/hypersensitivity or symptoms/signs of ongoing allergy/hypersensitivity
* Intake of any prescribed medicine or St John's Wort, except for occasional paracetamol and nasal anticongestant, within 3 weeks or use of over-the-counter drugs within 2 weeks before the first administration of study drug

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 112 (Actual)
Dates: Start 2007-11; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of AZD0328 by assessment of vital signs, laboratory variables and ECG | Assessments taken at visit 1 (enrolment), during visit 2 (residential period) and follow up visit 3.
Safety and tolerability of AZD0328 by assessment of adverse events | Non serious adverse events will be collected from the start of residential period until the end of the study. Serious adverse events will be collected from signing of consent until end of study.

SECONDARY OUTCOMES:
Determine the single and multiple dose pharmacokinetics (PK) of AZD0328 | PK sampling taken at defined timepoints during residential period.
Evaluate the cognitive dose response relationship for AZD0328 | Psychometric test battery performed at defined timepoints during residential period.

CONTACTS AND LOCATIONS:
Overall Officials: Wolfgang Kühn, Principal Investigator — Quintiles ABStrandbodgatan 1S-753 23 Uppsala; Erik Eliasson, MD, PhD, Study Chair — AstraZeneca R&D SödertäljeMedical Science S-151 85 Södertälje Sweden
Locations (4):
- Sweden (4):
  - Research Site, Linköping
  - Research Site, Luleå
  - Research Site, Stockholm
  - Research Site, Uppsala